CLINICAL TRIAL: NCT05978895
Title: FOOD-AUT Pilot Study Developing Canteen Menus Targeted to Nutritional and Sensory Needs of Adults With Autism Spectrum Disorder
Brief Title: FOOD-AUT Pilot Study Canteen Menus for Adults With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 30062023
Record Dates: First submitted 2023-07-19; First posted 2023-08-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; canteen menus; nutrition; food acceptance; sensory; color; texture; smell; sustainability; mealtime
MeSH Terms: conditions — Autism Spectrum Disorder; Anosmia

STUDY DESIGN:
Intervention Model Description: Non-randomized intervention with a single arm. Study participants received new adapted canteen menus according to the nutritional and sensory needs of the target population.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 22 adults with autism spectrum disorder (grade 1-2 or 3), admitted to the daycare service of Sacra Famiglia Onlus Foundation in Cesano Boscone (Milan, Italy)
  Interventions: Other: Targeted canteen menus

INTERVENTIONS:
Other: Targeted canteen menus — The nutritional intervention consisted in the development of targeted menus aiming at the needs of individuals with ASD and in assessing their acceptance of the targeted menus.
  The revision of the standard menus was carried 1) balancing energy and macronutrient content, according to LARN 2014; 2) promoting adequate weekly food frequencies consumption and portions, to provide an adequate and sustainable menus according to CREA 2018; 3) adapting the sensory characteristics of the foods offered to the sensory needs of individuals with ASD.
  The acceptance of the targeted menus by the enrolled population was evaluated through meal evaluation forms. These results were compared with the ones collected during the first observational phase (WP1). In fact, referring to the results of WP1, new canteen menus were drafted according to the nutritional and sensory needs of the population.

SUMMARY:
The FOOD-AUT pilot study aimed to improve the health status of adults with Autism Spectrum Disorder (ASD) through a nutritional intervention at canteen service. The researchers adapted the canteen menus to the nutritional and sensory needs of this vulnerable population, reducing their food selectivity and improving their dietary diversity with a positive impact on their health.

This project consisted of two phases: first an observational phase (Work Package 1, WP1) and secondarily an interventional phase (Work Package 2, WP2).

DETAILED DESCRIPTION:
The FOOD-AUT project was a pilot study conducted at the daycare service of Sacra Famiglia Onlus Foundation in Cesano Boscone (Milan, Italy) on adults with Autism Spectrum Disorder (ASD). The project lasted 12 months.

The main objective of the FOOD-AUT pilot study was to positively impact on the health condition of adults with ASD, improving food acceptability and increasing dietary diversity through the development of canteen service menus adapted to their nutritional and sensory needs.

The main outcome was the improvement of food acceptance of the canteen menus by the adults with ASD.

The FOOD-AUT pilot study deliverable were 1) the development of targeted canteen menus for adults with ASD, according to the nutritional and sensory needs; 2) the elaboration of dietary recommendations to customize canteen menus nutritional and sensory needs for individuals with ASD.

Participants of this study were adults (≥ 18 years old) diagnosed with an autism spectrum disorder (grade 1-2 or 3), admitted to the day care center for disabled persons (CDD) at Sacra Famiglia Fondazione Onlus (Cesano Boscone, Milan, Italy).

Based on the results of WP1, new canteen menus were drafted by qualified dietitians according to the nutritional and sensory needs of the targeted population. The new formulated menus 1) provided adequate caloric and macronutrient content, and 2) proposed with greater frequency foods having more accepted textures, colors, smells and temperatures.

A total of 12 meal evaluation forms for each participant were collected on 3 non-consecutive weekly days (for a total of 4 weeks). Both the qualitative and quantitative forms were filled out by qualified operators, previously trained, of the Sacra Famiglia Onlus Foundation, who assist the participants on a daily basis during lunches eaten at the facility. For the quantitative evaluation of food consumption, a score was assigned to the four possible amounts of dish consumed: zero consumption, ¼ of the plate, ½ of the plate, ¾ of the plate, the whole dish.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of autism spectrum disorder (grade 1-2 or grade 3)
* Admission to the daycare service of Sacra Famiglia Onlus Foundation in Cesano Boscone (Milan, Italy)
* Informed consent signed by their caregivers

Exclusion Criteria:

* Age < 18 years old
* Not diagnosed with autism spectrum disorder (grade 1-2 or grade 3)
* Not admitted to the daycare service of Sacra Famiglia Onlus Foundation in Cesano Boscone (Milan, Italy)
* Informed consent not signed by their caregivers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Food acceptance of canteen menus by adults with Autism Spectrum Disorder | 4 weeks (WP1); 4 weeks (WP2)
  Meal evaluation forms (score range for each item: 0-1; the score number is directly proportional to the amount of the dish consumed)

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, MD, Principal Investigator — University of Pavia
Locations (1):
- Sacra Famiglia, Cesano Boscone, Milan, Italy

REFERENCES:
- [Background] Conti MV, Breda C, Basilico S, Luzzi A, Voto L, Santero S, De Filippo G, Cena H. Dietary recommendations to customize canteen menus according to the nutritional and sensory needs of individuals with autism spectrum disorder. Eat Weight Disord. 2023 Aug 1;28(1):66. doi: 10.1007/s40519-023-01590-z. PMID 37526770
- [Derived] Conti MV, Santero S, Breda C, Basilico S, de Filippo G, Luzzi A, Voto L, Cavagnola R, Tomasinelli CE, Cena H. Autism Spectrum Disorder and collective catering service: results of the pilot study FOOD-AUT. Front Nutr. 2024 Jan 10;10:1298469. doi: 10.3389/fnut.2023.1298469. eCollection 2023. PMID 38268678